CLINICAL TRIAL: NCT01893905
Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of Chondroitin Sulfate and Glucosamine Sulfate in Combination Versus Placebo in Patients With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of a New Formulation of Chondroitin Sulfate and Glucosamine Sulfate to Treat Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tedec-Meiji Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TM-CS+SG /301; 2013-000444-26 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS+SG (Experimental): Chondroitin sulfate 1200mg+ glucosamine sulfate 1500mg orally administered once a day for 24 weeks
  Interventions: Drug: CS+SG
- Placebo (Placebo Comparator): Placebo of chondroitin sulfate + glucosamine sulfate orally administered once a day for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CS+SG — Chondroitin sulfate+glucosamine sulfate orally administered once a day for 24 weeks.
  Other Names: Chondroitin sulfate+glucosamine sulfate
  Arms: CS+SG
Drug: Placebo — Placebo of chondroitin sulfate+glucosamine sulfate orally administered once a day for 24 weeks.
  Other Names: Placebo chondroitin sulfate+glucosamine sulfate
  Arms: Placebo

SUMMARY:
The main objective is to assess the efficacy of a new formulation containing chondroitin sulfate and glucosamine sulfate (CS+GS) compared with placebo in patients with primary osteoarthritis of the knee.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a new combination of chondroitin sulfate and glucosamine sulfate administered once a day is superior to placebo in the treatment of patients with moderate to severe knee osteoarthritis. Eligible patients will be randomized 1:1 and the treatments will be administered for 24 weeks. Clinical efficacy at the end of treatment will be evaluated. Safety will be evaluated through adverse events recoding during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 45 years .
* Primary OA of the knee according to ACR criteria.
* OA radiological grade II-III according to Kellgren and Lawrence.
* Patients with moderate-severe pain.

Exclusion Criteria:

* Patients with clinical significant trauma or surgery in the target knee.
* Concurrent arthritic disease (antecedents and/or current signs) that could confound or interfere with the evaluation of pain efficacy such as chondrocalcinosis, Paget's disease of the ipsilateral limb to the target knee, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis, seronegative spondyloarthropathy, mixed connective tissue disease, collagen vascular disease, psoriasis, inflammatory bowel disease or fibromyalgia.
* Pain in other parts of the body greater than the knee pain that could interfere with the evaluation.
* Subjects with any active acute or chronic infections requiring antimicrobial therapy, or serious viral (e.g., hepatitis, herpes zoster, HIV positivity) or fungal infections.
* Clinical diagnosis established of uncontrolled diabetes mellitus.
* Patients with asthma.
* History of hypersensitivity to the active drugs or any excipients of the formulations.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FJ Blanco, M.D., Principal Investigator — Complejo Hospitalario Universitario La Coruña
Locations (1):
- Complejo Hospitalario Universitario La Coruña, A Coruña, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roman-Blas JA, Castaneda S, Sanchez-Pernaute O, Largo R, Herrero-Beaumont G; CS/GS Combined Therapy Study Group. Combined Treatment With Chondroitin Sulfate and Glucosamine Sulfate Shows No Superiority Over Placebo for Reduction of Joint Pain and Functional Impairment in Patients With Knee Osteoarthritis: A Six-Month Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Arthritis Rheumatol. 2017 Jan;69(1):77-85. doi: 10.1002/art.39819. PMID 27477804

RESULTS

PARTICIPANT FLOW:
Groups:
- CS+SG: Chondroitin sulfate+ glucosamine sulfate
- Placebo: Oral Placebo
Period: Overall Study
Arm/Group | CS+SG | Placebo
Started | 80 | 78
Completed | 55 | 64
Not Completed | 25 | 14
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 9 | 3
Not completed — Lack of Efficacy | 5 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 6 | 1
Not completed — Lack of adherence to treatment | 2 | 0
Not completed — Other reason | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- CS+SG: Chondroitin sulfate+glucosamine sulfate
- Placebo: Placebo oral
- Total: Total of all reporting groups
Arm/Group | CS+SG | Placebo | Total
Number analyzed (Participants) | 80 | 78 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.49 (8.17) | 67.60 (8.90) | 66.53 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 132
  Male | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain According to VAS (0-100 mm)
Description: VAS=The visual analogue scale is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, the patients specify their condition by indicating a position along a continuous line between two end-points. In our case a 0-100 mm line was used to define the degree of pain. The change between baseline and each evaluation visit (week 4, week 12 and week 24) was calculated to evaluate the efficacy of the treatments (a negative number represents a decrease in pain).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CS+SG | Placebo
Number analyzed (Participants) | 80 | 78
units on a scale | -11.86 (2.42) | -20.57 (2.41)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p < 0.0307, Pocock approach

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CS+SG | Placebo
Serious Adverse Events (participants affected / at risk) | 2/80 | 2/78
Other Adverse Events (participants affected / at risk) | 20/80 | 18/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CS+SG (N=80) | Placebo (N=78)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CS+SG (N=80) | Placebo (N=78)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No